CLINICAL TRIAL: NCT00497471
Title: The Prevention of Anaemia and Malaria in Infants in an Area of Intense and Perennial Malaria Transmission
Brief Title: RCT Iron Supplementation and Malaria Chemoprophylaxis for Prevention of Severe Anemia and Malaria in Tanzanian Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Follow-up end in 1999
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Agencia Española de Cooperación Internacional (Other); World Health Organization (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: IronMal
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-07

CONDITIONS: Malaria; Anemia
Keywords: Plasmodium Falciparum; Antimlarial chemoprophylaxis; Iron supplementation; Tanzania
MeSH Terms: conditions — Malaria; Anemia; Malaria, Falciparum | interventions — Pyrimethamine; Dapsone; Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Deltaprim (3.125 mg pyrimethamine plus 25 mg dapsone)
Drug: iron (2 mg/kg/daily)

SUMMARY:
The purpose of this trial is to evaluate the efficacy of weekly iron supplementation and the efficacy of malaria chemoprophylaxis from 2 to 12 months of age in infants living in an area of intense and perennial malaria transmission

DETAILED DESCRIPTION:
411 Tanzanian infants were randomly assigned to receive weekly malaria prophylaxis with Deltaprim™ (3.125 mg pyrimethamine plus 25 mg dapsone) or placebo from ages 2-12 months. Children were followed-up until age 4 years. Uncomplicated febrile malaria, severe malaria and anaemia morbidity were assessed through hospital-based passive surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Born in San Francis Designated District Hospital of Ifakara

Exclusion Criteria:

* Obvious severe congenital malformation such as: spina bifida, hydrocephalus or anencepahlus
* Twins
* Birth weight < 1,5 kg
* Clinical signs of cerebral asphyxia
* Clinical signs of neonatal or congenital infection
* Mother unreliable (deaf, mentally handicapped)

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 832 (Actual)
Dates: Start 1995-02; Study Completion 1999-07 (Actual)

PRIMARY OUTCOMES:
Clinical Malaria | During first year of life
Severe Anemia (PCV < 25%) | During first year of life

SECONDARY OUTCOMES:
Clinical Malaria | After first year of life
Severe Anemia (PCV < 25%) | After first year of life
Outpatient visits
Hospital Admissions
Severe malaria

CONTACTS AND LOCATIONS:
Overall Officials: Clara Menendez, MD, PhD, Principal Investigator — Centre for International Health, Hospital Clinic / Universitat Barcelona
Locations (1):
- Ifakara Centre, Ifakara, Tanzania

REFERENCES:
- [Result] Menendez C, Kahigwa E, Hirt R, Vounatsou P, Aponte JJ, Font F, Acosta CJ, Schellenberg DM, Galindo CM, Kimario J, Urassa H, Brabin B, Smith TA, Kitua AY, Tanner M, Alonso PL. Randomised placebo-controlled trial of iron supplementation and malaria chemoprophylaxis for prevention of severe anaemia and malaria in Tanzanian infants. Lancet. 1997 Sep 20;350(9081):844-50. doi: 10.1016/S0140-6736(97)04229-3. PMID 9310602